CLINICAL TRIAL: NCT00303303
Title: The Efficacy of Crotaline Fab Antivenom for Copperhead Snake Envenomations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to declining enrollment; data analysis proceeding.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-01-12B
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2013-08

CONDITIONS: Snake Envenomation
Keywords: Snake envenomation; Antivenins; Disability evaluation; Activities of daily living
MeSH Terms: conditions — Snake Bites | interventions — Red Meat; Maintenance; Crotalidae Polyvalent immune Fab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fab initial and maintenance therapy (Experimental): Active Fab Antivenom initial therapy followed by active Fab antivenom maintenance therapy
  Interventions: Biological: Crotaline Polyvalent Immune Fab (ovine) (active initial and maintenance therapy)
- Fab initial therapy; placebo maintenance (Experimental): Active initial Fab antivenom therapy followed by placebo maintenance therapy.
  Interventions: Biological: Crotaline Immune Fab (ovine) (active initial therapy; placebo maintenance therapy)
- Placebo initial and maintenance therapy (Placebo Comparator): Placebo initial and maintenance therapy.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Crotaline Polyvalent Immune Fab (ovine) (active initial and maintenance therapy) — Crotaline Polyvalent Immune Fab (Ovine), 4 vials initially; Second 4-vial dose two hours later if needed to achieve initial control of the envenomation syndrome; active maintenance therapy with 2 vials administered 6, 12, and 18 hours after initial control is achieved.
  Other Names: CroFab (tm)
  Arms: Fab initial and maintenance therapy
Biological: Crotaline Immune Fab (ovine) (active initial therapy; placebo maintenance therapy) — Crotaline Polyvalent Immune Fab (Ovine), 4 vials initially; Second 4-vial dose two hours later if needed to achieve initial control of the envenomation syndrome; placebo maintenance therapy administered 6, 12, and 18 hours after initial control is achieved.
  Other Names: CroFab (tm)
  Arms: Fab initial therapy; placebo maintenance
Biological: Placebo — Placebo therapy in place of initial and maintenance antivenom therapy. Note that open-label rescue therapy is mandated if the envenomation syndrome becomes severe, or if progression of envenomation signs/symptoms has not spontaneously halted by 6 hours.
  Arms: Placebo initial and maintenance therapy

SUMMARY:
Most patients bitten by copperhead snakes do not currently receive antivenom. Some snakebite victims have long term problems with the function of the limb that was bitten. This study will determine whether early administration of antivenom to patients with mild to moderate copperhead snakebites reduces long-term complications.

DETAILED DESCRIPTION:
This study seeks to answer three important questions about the role of ovine (sheep-derived) antivenom in the treatment of people bitten by copperhead snakes (Agkistrodon contortrix):

1. Although ovine antivenom has been approved by the FDA for treatment of copperhead envenomation, copperhead victims were excluded from the previous clinical trials. Animal experiments and retrospective human data suggest that the antivenom probably does work for copperhead snakebite, at least in the short term. This study will determine whether the antivenom is actually effective in reducing pain, swelling, and other immediate effects of copperhead snakebite.
2. Deaths from copperhead snakebite are extremely rare, but survivors often report long term problems with pain and swelling in the envenomated limb. No study has formally measured the long-term outcomes in untreated snakebite, nor whether antivenom has any benefit in reducing the duration or severity of these complications. This study will answer this question through formal assessments of limb function up to 12 months after treatment.
3. After initial control of the signs and symptoms of snakebite is achieved with antivenom therapy, some patients develop recurrent swelling or blood clotting problems. A randomized controlled trial in rattlesnake victims showed that the frequency of these problems is reduced by administration of 6 additional vials of antivenom over 18 hours ("maintenance therapy"). However, blood clotting problems are uncommon in copperhead snakebite even without antivenom treatment, and a retrospective trial suggested that maintenance therapy may have no effect on the frequency of delayed swelling in copperhead victims. In the typical copperhead victim, maintenance therapy increases the cost of treatment by more than 100%. This study will determine whether maintenance therapy is necessary in mild to moderate copperhead snakebite.

Patients are eligible for enrollment if they have been bitten by a snake positively identified as a copperhead within 6 hours of enrollment, if they have signs of mild or moderate severity envenomation, and if contraindications are not present.

After appropriate informed consent, patients are randomized to receive:

A. initial stabilizing dose of antivenom, followed by maintenance therapy,

B. initial stabilizing dose of antivenom followed by placebo in lieu of maintenance therapy, or

C. placebo for both initial dose and maintenance.

All laboratory testing, pain medication, hospitalization, and other therapies are standard for snakebite of this severity. If at any time the envenomation becomes severe, antivenom is administered.

In addition to the standard assessments performed on all snakebite victims (swelling, pain, vital signs, blood clotting, complications of therapy), patients in this study receive formal assessments of the function of the envenomated limb. This assessment uses the AMA disability rating system and the American Academy of Orthopedic Surgeons' Normative Outcomes Study questionnaire do determine how well the limbs function and how well the limbs perform and how much any remaining problems interfere with the patients' long-term happiness and ability to perform common activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Envenomation by copperhead snake (Agkistrodon contortrix) within 6 hours
* Mild or moderate severity envenomation

Exclusion Criteria:

* Allergy to antivenom or components
* Severe envenomation (hypotension, severe swelling, compartment syndrome, bleeding, etc.)
* Uncertain snake ID
* Prior treatment with antivenom

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P Kerns, MD, Principal Investigator — Carolinas Medical Center
Locations (4):
- United States (4):
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Richland Memorial Hospital, Columbia, South Carolina
  - Medical College of Virigina/Virginia Commonwealth University Hospital, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Fab Antivenom Followed by Fab Antivenom Maintenance: Fab Antivenom followed by Fab antivenom maintenance
- Fab Antivenom Followed by Placebo Maintenance Therapy: Fab antivenom followed by placebo maintenance therapy
- Placebo Initial Followed by Placebo Maintenance Therapy: Placebo initial and maintenance therapy
Period: Overall Study
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Started | 5 | 4 | 4
Completed | 5 | 4 | 3
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Fab Initial and Maintenance Therapy: Active Fab Antivenom initial therapy followed by active Fab antivenom maintenance therapy
- Experimental: Fab Initial Therapy; Placebo Maintenance: Active initial Fab antivenom therapy followed by placebo maintenance therapy.
- Placebo Comparator: Placebo Initial and Maintenance Therapy: Placebo initial and maintenance therapy.
- Total: Total of all reporting groups
Arm/Group | Experimental: Fab Initial and Maintenance Therapy | Experimental: Fab Initial Therapy; Placebo Maintenance | Placebo Comparator: Placebo Initial and Maintenance Therapy | Total
Number analyzed (Participants) | 5 | 4 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 4 | 4 | 4 | 12
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (19.9) | 41 (14.9) | 39 (19) | 38.2 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 1 | 3 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Limb Function: AMA Disability Rating Score of Envenomated Limb
Description: The range of possible scores is 0 - 100, and a lower score denotes less disability.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: Fab Antivenom followed by Fab antivenom maintenance
- Group 2: Fab antivenom followed by placebo maintenance therapy
- Group 3: Placebo initial and maintenance therapy
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 5 | 4 | 3
units on a scale | 11.2 (17.20) | 7.75 (7.18) | 22.67 (24.70)

2. Primary Outcome: Limb Function: AAOS Normative Outcome Study Scoring for Envenomated Limb
Description: Score ranges from 0-100 with higher scores meaning better function.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fab Initial and Maintenance Therapy | Fab Initial Therapy; Placebo Maintenance | Placebo Initial and Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
score on a scale | 48.4 (19.2) | 40.7 (14.7) | 40.3 (9.8)

3. Primary Outcome: Limb Function: AAOS Normative Outcome Study Scoring for Envenomated Limb
Description: Score ranges from 0-100 with higher scores meaning better function.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
score on a scale | 55.78 (2.45) | 55.18 (2.04) | 54.09 (3.96)

4. Primary Outcome: Limb Function: AAOS--time to Return to Normal Value
Description: Score ranges from 0-100 with higher scores meaning better function. Time in days to return to baseline value.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
days | 3.6 (2.8) | 5.5 (1.66) | 6.3 (1.70)

5. Secondary Outcome: Pain: Visual Analog Score
Description: 0-100 mm visual analog scale. Lower scores mean less pain.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
score on a scale | .5 (1.0) | 6.5 (7.3) | 19.0 (18.7)

6. Secondary Outcome: Pain Medication Use
Description: Mg of morphine equivalents
Time Frame: First 6 hours from baseline, first 18 hours from baseline, First 24 hours from baseline, 12 months
Population: Collected only for first 24 hours. Month 12 not collected.
Measure: Mean (Standard Deviation); unit: miligrams
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
miligrams
  First 24 hours from baseline | 5.2 (6.6) | 43.5 (40.5) | 29.9 (15.6)
  First 6 hours from baseline | 4.4 (4.45) | 15.95 (9.32) | 13.1 (2.45)
  first 18 hours from baseline | .8 (1.6) | 27.5 (28.9) | 16.8 (13.38)

7. Secondary Outcome: Swelling: Percentage (%) of Limb Spread Proximal From Bite Site
Time Frame: 12 months
Population: Data not collected
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Swelling: % Change in Volume Compared to Contralateral (Non-envenomated) Limb
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
percentage of change | 1 (5) | 2 (6) | -8 (9)

9. Secondary Outcome: Limb Function: Return to Work
Time Frame: Week 4
Population: At week 4: data not collected from 3 participants in Fab Antivenom followed by Fab antivenom maintenance arm; data not collected from 3 participants in the Fab antivenom followed by placebo maintenance therapy arm; no data collected in the Placebo initial followed by placebo maintenance therapy arm. Data not collected at month 12 for any participants
Measure: Median (Standard Deviation); unit: days
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 2 | 1 | 0
days | 3.75 (.25) | 4 |

10. Secondary Outcome: Limb Function: Physical or Occupational Therapy Sessions Attended
Time Frame: Week 4
Population: At week 4: data not collected from 3 participants in Fab Antivenom followed by Fab antivenom maintenance arm; data not collected from 3 participants in the Fab antivenom followed by placebo maintenance therapy arm; data only collected from 1 in the Placebo initial followed by placebo maintenance therapy arm. Data not collected at month 12 for any participants
Measure: Number; unit: number of sessions
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 2 | 1 | 1
number of sessions | 0 | 0 | 0

11. Secondary Outcome: Hematological: Clotting Studies and Platelet Counts
Time Frame: 12 months
Population: Data not collected at month 12
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Complications of Therapy
Description: Number of participants with acute hypersensitivity reactions
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fab Antivenom Followed by Fab Antivenom Maintenance | Fab Antivenom Followed by Placebo Maintenance Therapy | Placebo Initial Followed by Placebo Maintenance Therapy
Number analyzed (Participants) | 5 | 4 | 3
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 0/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=4) | Group 3 (N=4)
Acute hypersensitivity reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No